CLINICAL TRIAL: NCT01532973
Title: A Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-8742 in Hepatitis C Infected Males
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of Elbasvir (MK-8742) in Hepatitis C Infected Males (MK-8742-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8742-002; 2011-005190-23 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis, Viral, Human
MeSH Terms: conditions — Hepatitis, Viral, Human | interventions — elbasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- GT1 HCV 10-mg Elbasvir (Panel A) (Experimental): Participants with GT1 HCV receive 10 -mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GTI HCV 50-g Elbasvir (Panel B) (Experimental): Participants with GT1 HCV receive 50-mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT1 HCV 5-mg Elbavir (Panel C) (Experimental): Participants with GT1 HCV receive 5-mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT1 HCV 200-mg Elbasvir (Panel D) (Experimental): Participants with GT1 HCV receive 200-mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT3 HCV 10-mg Elbasvir (Panel E) (Experimental): Participants with GT3 HCV receive 10-mg elbasvir or matching placebo for 5 consecutive days during Part II of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT3 HCV 50-mg Elbasvir (Panel F) (Experimental): Participants with GT3 HCV receive 50-mg elbasvir or matching placebo for 5 consecutive days during Part II of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT3 HCV 100-mg Elbasvir (Panel G) (Experimental): Participants with GT3 HCV receive 100-mg elbasvir or matching placebo for 5 consecutive days during Part II of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT3 HCV 200-mg Elbasvir (Panel H) (Experimental): Participants with GT3 HCV receive 200-mg elbasvir or matching placebo for 5 consecutive days during Part II of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT1a HCV 10-mg Elbasvir (Panel I) (Experimental): Participants with GT1a only HCV receive 10-mg elbasvir or matching placebo for 5 consecutive days during Part III of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo
- GT1a HCV 50-mg Elbasvir (Panel J) (Experimental): Participants with GT1a only HCV receive 50-mg elbasvir or matching placebo for 5 consecutive days during Part III of the study.
  Interventions: Drug: Elbasvir; Drug: Placebo

INTERVENTIONS:
Drug: Elbasvir — Elbasvir was administered orally by tablet(s)
Drug: Placebo — Dose-matched placebo tablets were administered orally.

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics (PK) and pharmacodynamics of elbasvir (MK-8742) in Hepatitis C Virus (HCV)-infected participants. There will be 3 parts to this study; Part I will enroll only genotype (GT) 1 HCV-infected participants, Part II will enroll GT3 HCV-infected participants, and Part III will enroll only GT1a HCV-infected participants. All parts may run concurrently, or Parts II and III may be staggered.

Hypothesis (Part I): At a once-daily dose that is sufficiently safe and well tolerated in HCV-infected participants, elbasvir administered for 5 consecutive days has superior antiviral activity in GT1 HCV-infected participants compared to placebo, as measured by change from baseline in plasma HCV ribonucleic acid (RNA; log 10 copies/mL) at Day 5, 24-hour postdose timepoint. (a true mean viral RNA reduction of at least 3 log10 is anticipated).

Hypothesis (Part II): At a dose that is sufficiently safe in GT3 HCV-infected participants, the mean maximum reduction in HCV viral load is greater following multiple dose oral administration of elbasvir as compared to placebo.

Hypothesis (Part III): At a once-daily dose that is sufficiently safe and well tolerated in HCV-infected participants, elbasvir administered for 5 consecutive days has superior antiviral activity in GT1a HCV-infected participants compared to placebo, as measured by change from baseline in plasma HCV RNA (log 10 copies/mL) at Day 5, 24-hour postdose timepoint. (a true mean viral RNA reduction of at least 3 log10 is anticipated).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 to ≤ 37 kg/m^2
* Clinical diagnosis of chronic HCV infection defined by positive serology for HCV for at least 6 months and detectable HCV RNA in peripheral blood ≥105 IU/mL at screening
* Participant must be infected with HCV GT1a, GT1b, or GT 3

Exclusion Criteria:

* Co-infection with GT1 and GT3
* Estimated creatinine clearance of ≤70 mL/min based on the Cockcroft-Gault equation
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal (excepting HCV infection), cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic disease
* Positive Hepatitis B surface antigen at the pre-study (screening) visit
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy (screening) visit.
* Previous treatments (s) with nonstructural protein 5A (NS5A) inhibitors
* <4 weeks since administration of any experimental protease inhibitor
* Previous exposure to interferon-alpha and/or ribavirin within 3 month prior to the first dose of elbasvir in the study
* Clinical or laboratory evidence of advanced or decompensated liver disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2013-05-17 (Actual); Study Completion 2013-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Liu R, Curry S, McMonagle P, Yeh WW, Ludmerer SW, Jumes PA, Marshall WL, Kong S, Ingravallo P, Black S, Pak I, DiNubile MJ, Howe AY. Susceptibilities of genotype 1a, 1b, and 3 hepatitis C virus variants to the NS5A inhibitor elbasvir. Antimicrob Agents Chemother. 2015 Nov;59(11):6922-9. doi: 10.1128/AAC.01390-15. Epub 2015 Aug 24. PMID 26303801
- [Result] Yeh WW, Fraser IP, Jumes P, Petry A, Lepeleire I, Robberechts M, Reitmann C, Van Dyck K, Huang X, Guo Z, Panebianco D, Nachbar RB, O'Mara E, Wagner JA, Butterton JR, Dutko FJ, Moiseev V, Kobalava Z, Huser A, Visan S, Schwabe C, Gane E, Popa S, Ghicavii N, Uhle M, Wagner F. Antiviral Activity, Safety, and Tolerability of Multiple Ascending Doses of Elbasvir or Grazoprevir in Participants Infected With Hepatitis C Virus Genotype-1 or -3. Clin Ther. 2018 May;40(5):704-718.e6. doi: 10.1016/j.clinthera.2018.03.002. Epub 2018 Apr 25. PMID 29703432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 Panels (Panel D in Part 1 and Panel H in Part 2) were planned but not performed. No participants were enrolled in either of these panels.
Groups:
- GT1 HCV 10-mg Elbasvir (Panel A): Participants with genotype (GT) 1 hepatitis C virus (HCV) receive 10 -mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
- GT1 HCV 50-g Elbasvir (Panel B): Participants with GT1 HCV receive 50-mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
- GT1 HCV 5-mg Elbasvir (Panel C): Participants with GT1 HCV receive 5-mg elbasvir or matching placebo for 5 consecutive days during Part I of the study.
Period: Part 1
Arm/Group | GT1 HCV 10-mg Elbasvir (Panel A) | GT1 HCV 50-g Elbasvir (Panel B) | GT1 HCV 5-mg Elbasvir (Panel C) | GT1 HCV 200-mg Elbasvir (Panel D) | GT3 HCV 10-mg Elbasvir (Panel E) | GT3 HCV 50-mg Elbasvir (Panel F) | GT3 HCV 100-mg Elbasvir (Panel G) | GT3 HCV 200-mg Elbasvir (Panel H) | GT1a HCV 10-mg Elbasvir (Panel I) | GT1a HCV 50-mg Elbasvir (Panel J)
Started | 6 | 6 | 6 | 0 (Planned panel not performed. No participants were enrolled.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | GT1 HCV 10-mg Elbasvir (Panel A) | GT1 HCV 50-g Elbasvir (Panel B) | GT1 HCV 5-mg Elbasvir (Panel C) | GT1 HCV 200-mg Elbasvir (Panel D) | GT3 HCV 10-mg Elbasvir (Panel E) | GT3 HCV 50-mg Elbasvir (Panel F) | GT3 HCV 100-mg Elbasvir (Panel G) | GT3 HCV 200-mg Elbasvir (Panel H) | GT1a HCV 10-mg Elbasvir (Panel I) | GT1a HCV 50-mg Elbasvir (Panel J)
Started | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 (Planned panel not performed. No participants were enrolled.) | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3
Arm/Group | GT1 HCV 10-mg Elbasvir (Panel A) | GT1 HCV 50-g Elbasvir (Panel B) | GT1 HCV 5-mg Elbasvir (Panel C) | GT1 HCV 200-mg Elbasvir (Panel D) | GT3 HCV 10-mg Elbasvir (Panel E) | GT3 HCV 50-mg Elbasvir (Panel F) | GT3 HCV 100-mg Elbasvir (Panel G) | GT3 HCV 200-mg Elbasvir (Panel H) | GT1a HCV 10-mg Elbasvir (Panel I) | GT1a HCV 50-mg Elbasvir (Panel J)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug. Participants who received placebo in Part 1, 2, or 3 are grouped together regardless of HCV GT or randomly assigned panel. 2 Panels (Panel D in Part 1 and Panel H in Part 2) were planned but not performed. No participants were enrolled in either of these panels.
Groups:
- GT1 HCV 10-mg Elbasvir (Panel A): Participants with GT1 Hepatitis who received 10 -mg elbasvir for 5 consecutive days during Part I of the study.
- GT1 HCV 50-g Elbasvir (Panel B): Participants with GT1 HCV receive 50-mg elbasvir for 5 consecutive days during Part I of the study.
- GT1 HCV 5-mg Elbasvir (Panel C): Participants with GT1 HCV receive 5-mg elbasvir for 5 consecutive days during Part I of the study.
- GT3 HCV 10-mg Elbasvir (Panel E): Participants with GT3 HCV receive 10-mg elbasvir for 5 consecutive days during Part II of the study.
- GT3 HCV 50-mg Elbasvir (Panel F): Participants with GT3 HCV receive 50-mg elbasvir for 5 consecutive days during Part II of the study.
- GT3 HCV 100-mg Elbasvir (Panel G): Participants with GT3 HCV receive 100-mg elbasvir for 5 consecutive days during Part II of the study.
- GT1a HCV 10-mg Elbasvir (Panel I): Participants with GT1a only HCV receive 10-mg elbasvir for 5 consecutive days during Part III of the study.
- GT1a HCV 50-mg Elbasvir (Panel J): Participants with GT1a only HCV receive 50-mg elbasvir for 5 consecutive days during Part III of the study.
- Placebo: Participants with GT1, GT3 or GT1a HCV who received placebo in Parts I, II, or II of the study.
- Total: Total of all reporting groups
Arm/Group | GT1 HCV 10-mg Elbasvir (Panel A) | GT1 HCV 50-g Elbasvir (Panel B) | GT1 HCV 5-mg Elbasvir (Panel C) | GT3 HCV 10-mg Elbasvir (Panel E) | GT3 HCV 50-mg Elbasvir (Panel F) | GT3 HCV 100-mg Elbasvir (Panel G) | GT1a HCV 10-mg Elbasvir (Panel I) | GT1a HCV 50-mg Elbasvir (Panel J) | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.8) | 36.8 (6.9) | 51.6 (8.8) | 34.8 (6.4) | 35.8 (8.9) | 34.6 (6.8) | 51.0 (5.0) | 53.2 (11.6) | 47.8 (10.8) | 43.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction From Baseline in Log10 Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Day 5 - HCV GT1
Description: HCV RNA levels were assessed at baseline (predose on Day 1) and 24 hours postdose on Day 5 using the Roche TaqMan HCV 2.0 assay and transformed to Log10 values. The lower limits of quantification (LLOQ) and detection (LLD) were 25 and 9.3 IU/mL, respectively. Least squares means and confidence intervals obtained from the linear mixed model with log10 HCV RNA reduction as response and a fixed effect for treatment, time and treatment by time interaction.
Time Frame: Baseline (Predose on Day 1) and 24-hour post-dose on Day 5
Population: All participants who complied with the protocol sufficiently to ensure that data would likely exhibit the effects of treatment, according to the underlying scientific model and had available data from at least 1 treatment. Data for placebo were grouped together regardless of genotype or randomly assigned panel. Panel D was not conducted.
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/mL
Groups:
- GT1 HCV 10-mg Elbasvir (Panel A): Participants with GT1 Hepatitis receive 10 -mg elbasvir for 5 consecutive days during Part I of the study.
- Placebo: Participants with HCV GT1, GT3 or GT1a who received placebo during Parts I, II, or III of the study.
Arm/Group | GT1 HCV 10-mg Elbasvir (Panel A) | GT1 HCV 50-g Elbasvir (Panel B) | GT1 HCV 5-mg Elbasvir (Panel C) | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 8
IU/mL | 4.25 [3.80 to 4.71] | 4.40 [3.95 to 4.86] | 3.56 [3.10 to 4.02] | 0.00 [-0.37 to 0.36]
Statistical Analysis 1: Comparison: GT1 HCV 10-mg Elbasvir (Panel A) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 4.26, 90% CI 2-sided [3.77 to 4.74]
Statistical Analysis 2: Comparison: GT1 HCV 50-g Elbasvir (Panel B) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 4.41, 90% CI 2-sided [3.92 to 4.90]
Statistical Analysis 3: Comparison: GT1 HCV 5-mg Elbasvir (Panel C) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 3.56, 90% CI 2-sided [3.08 to 4.05]

2. Primary Outcome: Mean Reduction From Baseline in Log10 Plasma HCV RNA at Day 5 - HCV GT3
Description: as for outcome 1
Time Frame: Baseline (Predose on Day 1) and 24-hour post-dose on Day 5
Population: All participants who complied with the protocol sufficiently to ensure that data would likely exhibit the effects of treatment, according to the underlying scientific model and had available data from at least 1 treatment. Data for placebo were grouped together regardless of genotype or randomly assigned panel. Panel H was not conducted.
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GT3 HCV 10-mg Elbasvir (Panel E) | GT3 HCV 50-mg Elbasvir (Panel F) | GT3 HCV 100-mg Elbasvir (Panel G) | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 8
IU/mL | 1.01 [0.38 to 1.65] | 2.06 [1.43 to 2.70] | 2.72 [2.08 to 3.35] | 0.00 [-0.50 to 0.50]
Statistical Analysis 1: Comparison: GT3 HCV 10-mg Elbasvir (Panel E) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 1.02, 90% CI 2-sided [0.34 to 1.69]
Statistical Analysis 2: Comparison: GT3 HCV 50-mg Elbasvir (Panel F) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 2.07, 90% CI 2-sided [1.39 to 2.74]
Statistical Analysis 3: Comparison: GT3 HCV 100-mg Elbasvir (Panel G) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 2.72, 90% CI 2-sided [2.05 to 3.39]

3. Primary Outcome: Mean Reduction From Baseline in Log10 Plasma HCV RNA at Day 5 - HCV GT1a
Description: as for outcome 1
Time Frame: Baseline (Predose on Day 1) and 24-hour post-dose on Day 5
Population: All participants who complied with the protocol sufficiently to ensure that data would likely exhibit the effects of treatment, according to the underlying scientific model and had available data from at least 1 treatment. Data for placebo were grouped together regardless of genotype or randomly assigned panel.
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GT1a HCV 10-mg Elbasvir (Panel I) | GT1a HCV 50-mg Elbasvir (Panel J) | Placebo
Number analyzed (Participants) | 5 | 5 | 8
IU/mL | 3.20 [2.71 to 3.68] | 3.95 [3.46 to 4.43] | 0.00 [-0.39 to 0.38]
Statistical Analysis 1: Comparison: GT1a HCV 10-mg Elbasvir (Panel I) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 3.20, 90% CI 2-sided [2.68 to 3.72]
Statistical Analysis 2: Comparison: GT1a HCV 50-mg Elbasvir (Panel J) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 3.95, 90% CI 2-sided [3.44 to 4.47]

4. Primary Outcome: Mean Maximum Reduction in Log10 HCV Viral Load - HCV GT1
Description: HCV RNA levels were assessed at baseline (predose Day 1) and 24 hours postdose on Days 1-5. using the Roche TaqMan HCV 2.0 assay and transformed to Log10 values. The lower limits of quantification (LLOQ) and detection (LLD) were 25 and 9.3 IU/mL, respectively. The change in log10 LS mean HCV RNA levels was calculated for each timepoint and the maximum change from baseline was recorded.
Time Frame: Up to 5 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GT1 HCV 10-mg Elbasvir (Panel A) | GT1 HCV 50-g Elbasvir (Panel B) | GT1 HCV 5-mg Elbasvir (Panel C) | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 8
IU/mL | 4.44 [3.78 to 5.09] | 5.21 [4.56 to 5.87] | 4.15 [3.50 to 4.81] | 0.54 [0.03 to 1.06]
Statistical Analysis 1: Comparison: GT1 HCV 10-mg Elbasvir (Panel A) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 3.89, 90% CI 2-sided [3.20 to 4.58]
Statistical Analysis 2: Comparison: GT1 HCV 50-g Elbasvir (Panel B) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 4.67, 90% CI 2-sided [3.98 to 5.36]
Statistical Analysis 3: Comparison: GT1 HCV 5-mg Elbasvir (Panel C); Test type: Superiority or Other; Difference in LS Means = 3.61, 90% CI 2-sided [2.92 to 4.30]

5. Primary Outcome: Mean Maximum Reduction in Log10 HCV Viral Load - HCV GT3
Description: as for outcome 4
Time Frame: Up to 5 days
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GT3 HCV 10-mg Elbasvir (Panel E) | GT3 HCV 50-mg Elbasvir (Panel F) | GT3 HCV 100-mg Elbasvir (Panel G) | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 8
IU/mL | 1.27 [0.49 to 2.04] | 3.12 [2.34 to 3.89] | 3.38 [2.61 to 4.16] | 0.54 [-0.07 to 1.16]
Statistical Analysis 1: Comparison: GT3 HCV 10-mg Elbasvir (Panel E) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 0.72, 90% CI 2-sided [-0.09 to 1.54]
Statistical Analysis 2: Comparison: GT3 HCV 50-mg Elbasvir (Panel F) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 2.57, 90% CI 2-sided [1.75 to 3.39]
Statistical Analysis 3: Comparison: GT3 HCV 100-mg Elbasvir (Panel G) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 2.84, 90% CI 2-sided [2.02 to 3.66]

6. Primary Outcome: Mean Maximum Reduction in Log10 HCV Viral Load - HCV GT1a
Description: as for outcome 4
Time Frame: Up to 5 days
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GT1a HCV 10-mg Elbasvir (Panel I) | GT1a HCV 50-mg Elbasvir (Panel J) | Placebo
Number analyzed (Participants) | 5 | 5 | 8
IU/mL | 3.72 [3.12 to 4.31] | 4.17 [3.57 to 4.77] | 0.54 [0.07 to 1.02]
Statistical Analysis 1: Comparison: GT1a HCV 10-mg Elbasvir (Panel I) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 3.17, 90% CI 2-sided [2.55 to 3.80]
Statistical Analysis 2: Comparison: GT1a HCV 50-mg Elbasvir (Panel J) vs Placebo; Test type: Superiority or Other; Difference in LS Means = 3.63, 90% CI 2-sided [3.00 to 4.26]

7. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE) - Day 1 to Day 5
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE.
Time Frame: Up to 5 days
Population: All participants who received at least 1 dose of study drug. Events reported by drug taken at time of event and not by panel or genotype
Measure: Number; unit: Participants
Groups:
- 5-mg Elbasvir: Participants with HCV GT1 who received 5 -mg elbasvir
- 10-g Elbasvir: Participants with HCV GT1, GT3, or GT1a who received 10-mg elbasvir
- 50-mg Elbasvir: Participants with HCV GT1, GT3, or GT1a who received 50-mg elbasvir
- 100-mg Elbasvir: Participants with HCV GT3 who received 100-mg elbasvir
- Placebo: Participants with HCV GT1, GT3 or GT1a who received placebo during.
Arm/Group | 5-mg Elbasvir | 10-g Elbasvir | 50-mg Elbasvir | 100-mg Elbasvir | Placebo
Number analyzed (Participants) | 5 | 15 | 15 | 5 | 8
Participants | 4 | 6 | 7 | 1 | 4

8. Primary Outcome: Number of Participants Who Had Study Drug Discontinued Due to an Adverse Event
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Participants who had study drug discontinued due to an AE were recorded.
Time Frame: Up to 5 days
Population: All participants who received at least 1 dose of study drug. Event summarized by drug taken at time of event and not by panel or genotype
Measure: Number; unit: Participants
Arm/Group | 5-mg Elbasvir | 10-g Elbasvir | 50-mg Elbasvir | 100-mg Elbasvir | Placebo
Number analyzed (Participants) | 5 | 15 | 15 | 5 | 8
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Days 1 to 5 for each panel and then up to 56 days post last dose for follow-up period
Description: Adverse events are reported by drug taken at time of event for Days1-5 and not by panel or genotype. Adverse events for the post-study follow-up period (Days 6 to 61) are reported as 1 group regardless of genotype or study drug or dose received.
Groups:
- Post-Study: All participants who received 5, 10, 50, or 100 mg of elbasvir or placebo in treatment period of study
Arm/Group | 5-mg Elbasvir | 10-g Elbasvir | 50-mg Elbasvir | 100-mg Elbasvir | Placebo | Post-Study
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15 | 0/15 | 0/5 | 0/8 | 0/48
Other Adverse Events (participants affected / at risk) | 4/5 | 6/15 | 7/15 | 1/5 | 4/8 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-mg Elbasvir (N=5) | 10-g Elbasvir (N=15) | 50-mg Elbasvir (N=15) | 100-mg Elbasvir (N=5) | Placebo (N=8) | Post-Study (N=48)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (5) | 5 (6) | 1 (3) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.